CLINICAL TRIAL: NCT00341848
Title: Postpartum Uterine Regression
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902075; 02-E-N075
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-06-17 (Actual); Status verified 2019-06-13

CONDITIONS: Uterine Leiomyoma
Keywords: Apoptosis; Environment; Infection; Inflammation; Leiomyoma; Uterine Leiomyoma; Uterus
MeSH Terms: conditions — Myofibroma; Infections; Inflammation; Leiomyoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Uterine leiomyomas are the leading cause of hysterectomy in the United States, accounting for over 200,000 procedures each year. Most epidemiologic studies of uterine leiomyoma show that parity has a protective association with leiomyoma, but the mechanism is not known. Both epidemiologic data and data from an animal model indicate that the protective association is not an artifact resulting from reduced fertility among women with fibroids. We hypothesize that the process of uterine regression following delivery results in loss of small fibroids due to selective apoptosis of transformed cells and the extensive remodeling of the entire uterus.

DETAILED DESCRIPTION:
Background: Uterine leiomyomas are the leading cause of hysterectomy in the United States, accounting for over 200,000 procedures each year. Most epidemiologic studies of uterine leiomyoma show that parity has a protective association with leiomyoma, but the mechanism is not known. Both epidemiologic data and data from an animal model indicate that the protective association is not an artifact resulting from reduced fertility among women with fibroids. We hypothesize that the process of uterine regression following delivery results in loss of small fibroids due to selective apoptosis of transformed cells and the extensive remodeling of the entire uterus.

Study Objectives: Monitor fibroids during pregnancy and after postpartum uterine regression to assess any loss of fibroids and change in size of fibroids.

Methods: Add a postpartum ultrasound examination to an existing epidemiologic study of pregnant women. The parent study documents fibroid number, size, and location with a 7 week ultrasound examination. With the additional postpartum ultrasound proposed here, data on fibroid number, size, and location through pregnancy and postpartum uterine regression will be collected on approximately 400 women. A subsample of 30 women will also have an MRI after their postpartum ultrasound in order to evaluate the sensitivity of ultrasound imaging.

Significance: This study will provide the first data on fibroid change with parturition/postpartum uterine regression for a large sample of women. If small fibroids disappear during this time, it will document a process that results in "natural regression" of these tumors in premenopausal women. Insights from the biology of this process may be useful in developing treatment that could be used by nonpregnant women with fibroids to induce tumor regression.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants in the Right From The Start Study must be 18 years old or older, pregnant, enrolled by 10 weeks of gestation, planning to carry pregnancy to term, no plans to move before delivery, and English speaking. Those who are found to have fibroids at either their 7-week, or 22-week ultrasound examination are eligible for this further postpregnancy study.

A small substudy of 30 women having MRIs to evaluate the sensitivity of the ultrasound imaging will include only participants with a single fibroid found at the early pregnancy ultrasound.

EXCLUSION CRITERIA FOR MRI:

Exclusion criteria for the MRI are weight greater than 250 pounds, currently pregnant, metal of specific types in the body (an artificial hip, a clip for brain aneurysm, a medical implant in the ear, metal fragment in the eye, or a pacemaker), history of claustrophobia, previous severe reaction to MRI contrast, and chronic kidney disease. A severe reaction would consist of bronchospasm (shortness of breath/difficulty breathing) or shock (sudden loss of blood pressure). Risk is less than 1/100,000 with Gd based contrast material. Any potential subject with a history of kidney disease will be excluded from the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 374 (Actual)
Dates: Start 2001-12-06; Study Completion 2019-06-13

PRIMARY OUTCOMES:
Monitor fibroids

CONTACTS AND LOCATIONS:
Overall Officials: Donna D Baird, Ph.D., Principal Investigator — National Institute of Environmental Health Sciences (NIEHS)
Locations (1):
- NIEHS, Research Triangle Park, Research Triangle Park, North Carolina, United States

REFERENCES:
- [Background] Brett KM, Marsh JV, Madans JH. Epidemiology of hysterectomy in the United States: demographic and reproductive factors in a nationally representative sample. J Womens Health. 1997 Jun;6(3):309-16. doi: 10.1089/jwh.1997.6.309. PMID 9201665
- [Background] Cramer SF, Patel A. The frequency of uterine leiomyomas. Am J Clin Pathol. 1990 Oct;94(4):435-8. doi: 10.1093/ajcp/94.4.435. PMID 2220671
- [Background] Chen CR, Buck GM, Courey NG, Perez KM, Wactawski-Wende J. Risk factors for uterine fibroids among women undergoing tubal sterilization. Am J Epidemiol. 2001 Jan 1;153(1):20-6. doi: 10.1093/aje/153.1.20. PMID 11159141